CLINICAL TRIAL: NCT05983510
Title: Long Term Outcomes After Visceral Aortic Endarteriectomy for Coral Reef Lesion
Brief Title: Outcomes After Visceral Aortic Coral Reef Surgery
Status: Completed | Type: Observational
Sponsor: University Paul Sabatier of Toulouse (Other)
Responsible Party: Principal Investigator, Aurélien Hostalrich, MD,PhD Principal investigator, University Paul Sabatier of Toulouse
Other Study IDs: Long term Coral Reef
Record Dates: First submitted 2023-07-19; First posted 2023-08-09 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Aortic Coral Reef

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Aortic endarteriectomy — Thoraco-phreno-lumbotomy with thoracic aortic cross clamping Longitudinal aortotomy Endarteriectomy of the aorta Direct closure more or less bypass to the visceral arteries and downstream aorta reconstruction.

SUMMARY:
Coral reef aorta is defined by a calcified stenosis of the visceral aorta which can cause leg claudication, renal failure and visceral ischemia depending the type and localisation of the stenosis.

This pathology is rare and is usually treated by open surgery with aortic endarteriectomy. Little is know about the outcomes after such aggressive surgery with short series and short follow up.

The authors propose a retrospective study from their institution to explore the post operative and long term outcomes after this surgery.

DETAILED DESCRIPTION:
Coral reef aorta is defined by a calcified stenosis of the visceral aorta which can cause leg claudication, renal failure and visceral ischemia depending the type and localisation of the stenosis.

This pathology is rare and is usually treated by open surgery with aortic endarteriectomy.

Little is known in the literature regarding the outcomes of this aggressive surgery.

The authors propose a retrospective study from their institution describing the type of surgery realised. They describe the post operative outcomes of this surgery in term of cardiologic, respiratory, renal complication a,d surgical complication.

Moreover they follow the patients to present long term outcomes of this pathology with a description of the post operative recurrence of a coral reef, the permeability of the different target vessel and the cardiologic, respiratory and renal evolution of the different patients.

ELIGIBILITY:
Inclusion Criteria:

* Coral reef surgery
* Urgent intervention
* Claudication, renal, visceral involvement
* Thoracic aortic cross clamping (above coeliac trunk)

Exclusion Criteria:

* "simple" visceral aorto thrombectomy without opening laterally the aorta
* Pregnant

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who needed a coral reef surgery were included
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac event (MACE) | 1 month after surgery
  Post operative cardiologic complication
Reintervention | 1 month after surgery
  Need of reintervention before discharge

SECONDARY OUTCOMES:
Long term follow up | 1 month, 1 year, yearly up to 5 years
  Cumulative survival rate
Target vessel patency | 1 month, 1 year, yearly up to 5 years
  Permeability of the different vessel (renal and visceral arteries) on CT scan or Duplex ultrasound
Kidney function evolution | 1 month, 1 year, yearly up to 5 years
  glomerular filtration rate evolution,

CONTACTS AND LOCATIONS:
Locations (1):
- Hostalrich Aurélien, Toulouse, France